CLINICAL TRIAL: NCT03067363
Title: Assessment of Safety, Tolerability and Pharmacokinetics of Single Ascending Subcutaneous Doses of MOR107 in Healthy Male Subjects and Pharmacodynamics in Healthy Male Subjects on a Low Sodium Diet
Brief Title: First in Human Single Ascending Dose Study of MOR107
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Part 1 completed successfully. Part 2 not conducted.
Sponsor: Alan Richardson (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor-Investigator, Alan Richardson, Clinical Project Manager, LanthioPep BV
Organization: LanthioPep BV (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MOR107-C001
Record Dates: First submitted 2017-02-21; First posted 2017-03-01 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Safety
MeSH Terms: interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Intervention Model Description: Part 1: single ascending doses Part 2: parallel group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Part 1, MOR107 Dose level 1 (Experimental): MOR107, single subcutaneous injection
  Interventions: Drug: MOR107
- Part 1, MOR107 Dose level 2 (Experimental): MOR107, single subcutaneous injection
  Interventions: Drug: MOR107
- Part 1, MOR107 Dose level 3 (Experimental): MOR107, single subcutaneous injection
  Interventions: Drug: MOR107
- Part 1, MOR107 Dose level 4 (Experimental): MOR107, single subcutaneous injection
  Interventions: Drug: MOR107
- Part 1, MOR107 Dose level 5 (Experimental): MOR107, single subcutaneous injection
  Interventions: Drug: MOR107
- Part 1, MOR107 Dose level 6 (Experimental): MOR107, single subcutaneous injection
  Interventions: Drug: MOR107
- Part 1, Placebo (Placebo Comparator): Placebo, single subcutaneous injection
  Interventions: Drug: Placebo
- Part 2: MOR107 low dose (Experimental): MOR107 low dose single subcutaneous injection and low sodium diet for 6 days before dosing and 2 days after dosing
  Interventions: Drug: MOR107; Other: Low sodium diet
- Part 2: MOR107 medium dose (Experimental): MOR107 medium dose single subcutaneous injection and low sodium diet for 6 days before dosing and 2 days after dosing
  Interventions: Drug: MOR107; Other: Low sodium diet
- Part 2: MOR107 high dose (Experimental): MOR107 high dose single subcutaneous injection and low sodium diet for 6 days before dosing and 2 days after dosing
  Interventions: Drug: MOR107; Other: Low sodium diet
- Part 2: Placebo (Placebo Comparator): Placebo single subcutaneous injection and low sodium diet for 6 days before dosing and 2 days after dosing
  Interventions: Drug: Placebo; Other: Low sodium diet

INTERVENTIONS:
Drug: MOR107 — MOR107 solution for injection
  Other Names: LP2-3
  Arms: Part 1, MOR107 Dose level 1; Part 1, MOR107 Dose level 2; Part 1, MOR107 Dose level 3; Part 1, MOR107 Dose level 4; Part 1, MOR107 Dose level 5; Part 1, MOR107 Dose level 6; Part 2: MOR107 high dose; Part 2: MOR107 low dose; Part 2: MOR107 medium dose
Drug: Placebo — Solution for injection manufactured to match MOR107 solution for injection
  Other Names: Placebo (for MOR107)
  Arms: Part 1, Placebo; Part 2: Placebo
Other: Low sodium diet — Diet designed to restrict sodium intake to 40 mmol/day
  Arms: Part 2: MOR107 high dose; Part 2: MOR107 low dose; Part 2: MOR107 medium dose; Part 2: Placebo

SUMMARY:
This is the first in human study of MOR107. It is a 2 part, single centre, double-blind, randomised, placebo-controlled study in healthy male subjects. Part 1 is a single ascending dose study, and Part 2 is a parallel group, dose range finding study in healthy male subjects on a low sodium diet.

DETAILED DESCRIPTION:
MOR107 is an angiotensin 2 receptor (AT2R) agonist with the potential to treat a wide range of diseases through activation of the protective arm of the renin-angiotensin system.

In this study MOR107 will be administered to humans for the first time.

The study will enroll healthy male subjects and is split into two sequential parts, both of which have a single centre, double-blind, randomised, placebo-controlled design.

Part 1 will evaluate the safety, tolerability and pharmacokinetics (PK) of single ascending doses of MOR107.

Part 2 will evaluate the pharmacodynamics, safety, tolerability and PK of three different doses of MOR107 in healthy male subjects who will be fed a low sodium diet in order to increase AT2R expression.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy males
2. Age 18 to 45 years of age
3. Body mass index of 18.0 to 32.0 kg/m2
4. For Part 2, subjects must have at least a 25% reduction in 24 hour urinary sodium excretion on Day -2 compared with admission

Key Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the previous three months
2. Regular alcohol consumption >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
3. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening/admission
4. Current smokers of e-cigarettes and nicotine replacement products and those who have smoked these products within the last 12 months
5. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator
6. Positive drugs of abuse test result
7. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
8. History of psychiatric disorder, cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease as judged by the investigator
9. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability) | Up to 10 days post-dose
  Reporting of adverse events, physical examination, injection site assessment, vital signs, ECG, and clinical chemistry, haematology and urinalysis

SECONDARY OUTCOMES:
Time from dosing at which the maximum MOR107 concentration was observed (Tmax) | Up to 48 hours post-dose
  Plasma PK parameter
Maximum observed MOR107 concentration (Cmax) | Up to 48 hours post-dose
  Plasma PK parameter
Concentration of MOR107 at 12 hours post-dose (C12) | 12 hours post-dose
  Plasma PK parameter
Concentration of MOR107 at 24 hours post-dose (C24) | 24 hours post-dose
  Plasma PK parameter
Area under the curve from 0 time to last measurable MOR107 concentration (AUC0-t) | Up to 48 hours post-dose
  Plasma PK parameter
Area under the curve from 0 time to infinity for MOR107 (AUC0-inf) | Up to 48 hours post-dose
  Plasma PK parameter
Percentage of AUC(0-inf) for MOR107 extrapolated beyond last measured time point (AUC%extrap) | Up to 48 hours post-dose
  Plasma PK parameter
Slope of the apparent elimination phase for MOR107 (Lambda-z) | Up to 48 hours post-dose
  Plasma PK parameter
Apparent elimination half-life for MOR107 (T-half) | Up 48 hours post-dose
  Plasma PK parameter
MOR107 Cmax normalised for dose (Cmax/D) | Up to 48 hours post-dose
  Plasma PK parameter
MOR107 AUC(0-t) normalised for dose (AUC[0-t]/D) | Up to 48 hours post-dose
  Plasma PK parameter
MOR107 AUC(0-inf) normalised for dose (AUC[0-inf]/D) | Up to 48 hours post-dose
  Plasma PK parameter
Amount of MOR107 excreted in the urine over a specified period of time after dosing (Ae) | Up to 48 hours post-dose
  Urine PK parameter
Cumulative amount of MOR107 excreted in the urine (CumAe) | Up to 48 hours post-dose
  Urine PK parameter
Amount of MOR107 excreted in the urine over a specified period of time after dosing, expressed as a percentage of the administered dose (Ae%) | Up to 48 hours post-dose
  Urine PK parameter
Cumulative amount of MOR107 excreted in the urine, expressed as a percentage of the administered dose (CumAe%) | Up to 48 hours post-dose
  Urine PK parameter
Renal clearance: the apparent volume of plasma cleared per unit time via renal elimination (CLr) | Up to 48 hours post-dose
  Urine PK parameter

CONTACTS AND LOCATIONS:
Overall Officials: Axel Mescheder, MD, Study Director — LanthioPep BV
Locations (1):
- Quotient Clinical, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No